CLINICAL TRIAL: NCT03765840
Title: Relationship Between Postoperative Cognitive Decline and Cytokines in Elderly Patients
Brief Title: Study of Postoperative Cognitive Decline in Aged Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jia-feng Wang (Other)
Responsible Party: Sponsor-Investigator, Jia-feng Wang, M.D, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: POCD-aged
Record Dates: First submitted 2018-12-02; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood of patients is collected preoperation and 24h after surgery and 72h after surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POCD group: patients occur cognitive decline after surgery according to scores in this group.
- NO POCD group: patients do not occur cognitive decline after surgery according to scores in this group.

SUMMARY:
postoperative cognitive decline is a common and deleterious complication in aged patients.The link between inflammation and postoperative cognitive decline has also been reported.However,the link between SOD1，SOD2，Osteopontin， Kallikrein-6，and Contactin-1 and postoperative cognitive decline is unknown. In this project ,investigators examine the relationship between 5 cytokines measured at there timepoints (preoperative [PREOP], postoperative day 1 [POD1] , and postoperative day 3[POD2]) and postoperative cognitive decline among older adults undergoing orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who are more than 65 years old
* patients who undergo orthopedic surgery(trauma ,especially fracture of lower limb)
* patients with ASA physical status I-III
* patients who have a consent

Exclusion Criteria:

* patients who are more than 85 years old
* patients with ASA physical status >III
* patients who have neurological disorders, stroke or other affective central nervous system diseases
* patients who have a history of serious psychiatric illness
* patients with long-term use of psychoactive substances
* patients who undergo multiple trauma and the presence of head injury

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: aged patients who recieve surgery for orthopedic surgery under spinal or general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Differences in cytokines levels between the two groups | preoperation
  Compare differences in cytokines levels between the two groups
Differences in cytokines levels between the two groups | 24h after operation
  Compare differences in cytokines levels between the two groups
Differences in cytokines levels between the two groups | 72h after operation
  Compare differences in cytokines levels between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Deartment of anesthesiology,changhai hospital, Shanghai, Shanghai Municipality, China